CLINICAL TRIAL: NCT04779034
Title: The Relationship Between Heart Rate Variation and Athletic Performance in Basketball Players
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ankara Yildirim Beyazıt University (Other)
Responsible Party: Principal Investigator, Rabia Tugba Kilic, assistant professor, Ankara Yildirim Beyazıt University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: AYBU195320103
Record Dates: First submitted 2021-01-28; First posted 2021-03-03 (Actual); Last update posted 2021-08-10 (Actual); Status verified 2021-02

CONDITIONS: Heart Rate Variability; Athletic Performance
Keywords: heart rate variability; athletic performance

STUDY DESIGN:
Intervention Model Description: to explain the relationship between heart rate variability and their sportive performance in basketball players.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Group 1 (Experimental): Basketball players
  Interventions: Other: Measurement of heart rate variability

INTERVENTIONS:
Other: Measurement of heart rate variability — Heart rate variation will be evaluated with the Polar RS800CX model heart rate monitor
  Other Names: demographic information; YoYo intermittent loading test; 20-meter speed test; vertical jump test; illionis agility test; lower extremity y balance test; upper extremity y balance test; medicine ball launch test; basketball-specific sports performances in shooting, passing, defense and dribbling tests

SUMMARY:
This study was planned to explain the relationship between heart rate variability and their sportive performance in basketball players.

DETAILED DESCRIPTION:
Basketball is a team sport that develops physical characteristics such as endurance, strength, speed, skill and mobility, starting from childhood or youth and bringing these characteristics to a superior level in adulthood.

The heart rate variability is the period in which the change between two heartbeats is observed and represents the sinus node modulation by the sympathetic and parasympathetic branches of the autonomic nervous system. During exercise, the increase in intensity produces a higher heart rate and a lower heart rate variation due to the increase in sympathetic nerve activity and decreased vagal modulation in the heart. Heart rate variation is measured by the variation in heart rate from beat to beat and the time between each heartbeat. Measurement of heart rate variability is a potentially valuable noninvasive tool as it is a reliable marker of the autonomic nervous system's effect on the heart.

When the literature is examined, although there are studies on the effects of heart rate variation in both basketball and different sports branches, there is no study examining the relationship between heart rate variation and basketball-specific sportive performance. Therefore, it is aimed to study on this subject and to contribute to the literature.

ELIGIBILITY:
Inclusion Criteria:

1. without any known systemic problems
2. without any history of musculoskeletal injuries in the last 6 months
3. men basketball player

Exclusion Criteria:

1. those who do not volunteer to participate

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 100 (Estimated)
Dates: Start 2021-08-01 (Estimated); Primary Completion 2021-10-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
Heart rate variability | 5 months
  Heart rate variability

SECONDARY OUTCOMES:
Athletic performance 1 | 5 months
  YoYo intermittent loading test
Athletic performance 2 | 5 months
  20-meter speed test
Athletic performance 3 | 5 months
  vertical jump test
Athletic performance 4 | 5 months
  illionis agility test
Athletic performance 5 | 5 months
  lower extremity y balance test
Athletic performance 6 | 5 months
  upper extremity y balance test
Athletic performance 7 | 5 months
  medicine ball launch test
Athletic performance 8 | 5 months
  shooting test
Athletic performance 9 | 5 months
  passing test
Athletic performance 10 | 5 months
  defense test
Athletic performance 11 | 5 months
  dribbling test

CONTACTS AND LOCATIONS:
Overall Officials: Burak Karahan, Study Chair — burakkarahan10@gmail.com
Locations (1):
- Ankara Yildirim Beyazit University,Faculty of Health Sciences, Physiotherapy and Rehabilitation Department, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ramos-Campo DJ, Rubio-Arias JA, Avila-Gandia V, Marin-Pagan C, Luque A, Alcaraz PE. Heart rate variability to assess ventilatory thresholds in professional basketball players. J Sport Health Sci. 2017 Dec;6(4):468-473. doi: 10.1016/j.jshs.2016.01.002. Epub 2016 Jan 12. PMID 30356606
- [Result] Prinsloo GE, Rauch HG, Derman WE. A brief review and clinical application of heart rate variability biofeedback in sports, exercise, and rehabilitation medicine. Phys Sportsmed. 2014 May;42(2):88-99. doi: 10.3810/psm.2014.05.2061. PMID 24875976
- [Result] Buckthorpe M, Morris J, Folland JP. Validity of vertical jump measurement devices. J Sports Sci. 2012;30(1):63-9. doi: 10.1080/02640414.2011.624539. Epub 2011 Nov 23. PMID 22111944